CLINICAL TRIAL: NCT04255602
Title: A Randomized Non-inferiority Study of Low-dose and Standard-dose Ticagrelor After Intervention for Acute Coronary Syndrome
Brief Title: A Study of Low and Standard-dose Ticagrelor After Intervention for ACS Patients
Acronym: TIGER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Tong Ren Hospital (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other); Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP2020125
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-10

CONDITIONS: Acute Coronary Syndrome; Coronary Stent Implantation
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low dose ticagrelor (Experimental): After treated with ticagrelor 90mg twice daily and aspirin 100mg once daily for a week,subjects will be treated with ticagrelor 60mg twice daily and aspirin 100mg once daily for until one year after drug eluting stent implantation
  Interventions: Drug: Ticagrelor 60mg
- standard dose ticagrelor (Active Comparator): subjects will be treated with ticagrelor 90mg twice daily and aspirin 100mg once daily for a year since drug eluting stent implantation
  Interventions: Drug: Ticagrelor 90mg

INTERVENTIONS:
Drug: Ticagrelor 60mg — Ticagrelor 60mg plus Aspirin 100mg for experimental group
  Arms: low dose ticagrelor
Drug: Ticagrelor 90mg — Ticagrelor 90mg plus Aspirin 100mg for active comparator group
  Arms: standard dose ticagrelor

SUMMARY:
This study is to evaluate the safety and efficacy of 60mg ticagrelor plus 100mg Aspirin to prevent major adverse cardiovascular and cerebrovascular events in one years after drug-eluting stents implantation for Chinese ACS patients compared with 90mg ticagrelor plus 100mg Aspirin

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age
2. Patients should have undergone successful percutaneous coronary intervention with drug-eluting stent for acute coronary syndrome
3. Subject understand the study requirements and the treatment procedures and provided informed consent before the procedure

Exclusion Criteria:

1. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study
2. Active bleeding
3. Known hypersensitivity or contraindication to study medications
4. Non-cardiac co-morbid conditions are present with life expectancy <2 year or that may result in protocol non-compliance (per site investigator's medical judgment).
5. Subjects with Cerebral hemorrhage history
6. Subjects with stroke history in half a year
7. subjects with malignant tumor
8. subjects with whom oral anticoagulants are needed

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2120 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
a composite of cardiovascular death, non-fatal myocardial infarction, stent thrombosis,coronary revascularization,stroke, and bleeding events of BARC grade ≥2 | Stent implantation to 12 months
  a composite of death from coronary vascular causes,non-fatal myocardial infarction,stent thrombosis,coronary revascularization, stroke and bleeding type 2, 3 or 5 according to the Bleeding Academic Research Consortium (BARC) criteria

SECONDARY OUTCOMES:
bleeding events of BARC grade ≥2 | Stent implantation to 12 months
  bleeding type 2, 3 or 5 according to the Bleeding Academic Research Consortium (BARC) criteria
a composite of cardiovascular death, non-fatal myocardial infarction, stent thrombosis,coronary revascularization,stroke | Stent implantation to 12 months
  a composite of cardiovascular death, non-fatal myocardial infarction, stent thrombosis,coronary revascularization,stroke

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Doctor, Study Chair — Fudan University; Lei Hou, Doctor, Principal Investigator — Shanghai Tongren Hospital
Locations (8):
- China (8):
  - Taishan people's hospital, Taishan, Guangdong
  - South East of Shandong hospital, Liaocheng, Shandong
  - zhangshan hospital, Fudan University, Shanghai, Shanghai Municipality
  - shanghai Tongren hospital, Shanghai, Shanghai Municipality
  - Minhang hospital, Fudan University, Shanghai, Shanghai Municipality
  - Songjiang hospital, Shanghai jiaotong university, school of medicine, Shanghai, Shanghai Municipality
  - Ningbo 4th hospital, Xiangshan, Zhejiang
  - Yanzhou branch of affiliated hospital of Jining medical university, Jining

REFERENCES:
- [Derived] Pang Y, Ma M, Xia J, Wang D, YanChen, Ye J, Jia Z, Wu S, Yang J, Hou L. A randomized non-inferiority study of low-dose and standard-dose ticagrelor after intervention for acute coronary syndrome: study protocol for the TIGER STUDY. Trials. 2022 Mar 5;23(1):203. doi: 10.1186/s13063-022-06124-z. PMID 35248132